CLINICAL TRIAL: NCT06402344
Title: Association of Hormonal Implant With Gestrinone on Endothelial Function in Young Women
Brief Title: Gestrinone and Endothelial Function in Young Women
Status: Recruiting | Type: Observational
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Sponsor
Other Study IDs: 75851223.3.0000.0071
Record Dates: First submitted 2024-04-26; First posted 2024-05-07 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2024-04

CONDITIONS: Cardiovascular Diseases
Keywords: Hormonal implant; Gestrinone; Endothelial function
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Control Groups

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gestrinone implant: Young women using hormonal implant with gestrinone.
  Interventions: Other: Hormonal implant
- Control group: Young women who never used hormonal implant with gestrinone.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Hormonal implant — History of at least 1 hormonal implant with gestrinone in the last 6 months, applied by the participant's private doctor.
  Groups: Gestrinone implant
Other: Control group — Young women who never used any hormonal implant.
  Groups: Control group

SUMMARY:
The purpose of this study is to assess the association of hormonal implant with gestrinone in cardiovascular health outcomes in young women.

DETAILED DESCRIPTION:
After being informed about the study, volunteers will be screened in accordance with eligibility criteria. Eligible volunteers will be invited to appear to the research institute and participate in the study. All volunteers giving the written informed consent will perform all assessments in the same day at their visit.

ELIGIBILITY:
Inclusion Criteria:

* Women;
* Between 25 and 45 years age;
* History of ≥ 1 hormonal implant with gestrinone in the last 6 months or never had used any hormonal implants.

Exclusion Criteria:

* Pregnancy;
* Menopause;
* Smoking;
* Moderate-high consumption of alcoholic beverages (above 14 drinks per week);
* Previous cardiovascular event (e.g. myocardial infarction and stroke);
* Uncontrolled psychiatric disease;
* Ventricular arrhythmia;
* Using antibiotics or corticoids;
* Regular contraceptive use (estrogen and progesterone);
* Use of illicit drugs.

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Young women.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-08-22 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Endothelial function | Day 1.
  Brachial artery endothelial function assessed by flow-mediated dilation (FMD).

SECONDARY OUTCOMES:
Arterial stiffness | Day 1.
  Carotid-femoral pulse wave velocity (PWV).
Heart rate | Day 1.
  Heart rate assessed together with the cardiac autonomic modulation procedure.
Blood pressure | Day 1.
  Systolic, diastolic and mean blood pressure will be evaluated by auscultatory method.
Cardiac autonomic modulation | Day 1.
  Heart rate variability (HRV) analyzed in the time domain, frequency domain, and non-linear method.
Lipid profile | Day 1.
  Total cholesterol, non-HDL cholesterol, low-density lipoprotein (LDL-c), high-density lipoprotein (HDL-c), and triglycerides will be analyzed by laboratory exams.
Glycemia | Day 1.
  Glycemia will be analyzed by laboratory exams.
Ultra-sensitive C-reactive protein (us-CRP) | Day 1.
  us-CRP will be analyzed by laboratory exams.
Hemoglobin | Day 1.
  Hemoglobin will be analyzed by laboratory exams.
Hematocrit | Day 1.
  Hematocrit will be analyzed by laboratory exams.
Progesterone | Day 1.
  Progesterone will be analyzed by immunoassay technique.
17-alpha-hydroxyprogesterone (17-OHP) | Day 1.
  17-OHP will be analyzed by liquid chromatography-mass spectrometry (LC-MS/MS).
Dehydroepiandrosterone (DHEA) | Day 1.
  DHEA will be analyzed by liquid chromatography-mass spectrometry (LC-MS/MS).
Androstenedione | Day 1.
  Androstenedione will be analyzed by liquid chromatography-mass spectrometry (LC-MS/MS).
Free testosterone | Day 1.
  Free testosterone will be calculated considering total testosterone and SHBG.
Total testosterone | Day 1.
  Total testosterone will be analyzed by liquid chromatography-mass spectrometry (LC-MS/MS).
Estradiol | Day 1.
  Estradiol will be analyzed by immunoassay technique.
Follicle-stimulating hormone (FSH) | Day 1.
  FSH will be analyzed by immunoassay technique.
Luteinizing hormone (LH) | Day 1.
  LH will be analyzed by immunoassay technique.
Sex hormone-binding globulin (SHBG) | Day 1.
  SHBG will be analyzed by immunoassay technique.
Muscular strength | Day 1.
  It will be assessed by handgrip.

CONTACTS AND LOCATIONS:
Overall Officials: Luciana Diniz Nagem Janot de Matos, MD, PhD, Principal Investigator — Medical Referencee - Rehabilitation Center
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
There will be no individual participant data (IPD) shared.